CLINICAL TRIAL: NCT03153878
Title: The Prospective Cohort Study on the Benefit-risk of Antithrombotic or Anticoagulant Therapy in Patients With Unruptured Intracranial Aneurysms Associated With Ischemic Heart Disease or Ischemic Cerebrovascular Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Liu Zhiyong (Other)
Collaborators: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor-Investigator, Liu Zhiyong, Research associate, West China Hospital
Organization: West China Hospital (Other)
Other Study IDs: 2016YFC1300803
Record Dates: First submitted 2017-05-11; First posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Intracranial Aneurysm; Natural History; Ischemic Heart Disease; Ischemic Cerebrovascular Disease
Keywords: Unruptured Intracranial Aneurysm; Benefit-risk; Ischemic heart disease; Ischemic cerebrovascular disease; Antithrombotic; Anticoagulant; People's Republic of China; Multicenter Studies
MeSH Terms: conditions — Intracranial Aneurysm; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a registry study of the natural course of unruptured intracranial aneurysms (UIA). In addition, the investigators will analyze the benefit-risk of antithrombotic or anticoagulant therapy in patients with unruptured intracranial aneurysms associated with ischemic heart disease or ischemic cerebrovascular disease. The investigators aim to use research data to create a China national database of UIA

DETAILED DESCRIPTION:
This is a registry study of the natural course of unruptured intracranial aneurysms (UIA). In addition, the investigators will analyze the benefit-risk of antithrombotic or anticoagulant therapy in patients with unruptured intracranial aneurysms associated with ischemic heart disease or ischemic cerebrovascular disease. The investigators aim to use research data to create a China national database of UIA. This study is supported by a research grant from the Ministry of Science and Technology of the People's Republic of China. The investigators will collaborate with the other 19 medical centers which locate in the different districts of China.

During the study period, all the patients included in this study will observe and treat in the collaborating medical centers. Included patients will be followed-up for at least 1year. Research data will represent the real natural course of UIA in China. For this study, the investigators consulted and hired professional experts about data collection, data and methodology. An intact systematic project steering committee, including Data Monitoring Committee, Data Management Committee, Project Academic Committee, Executive Group, Project Manager, Project Statistician, and Technical Support Center has been built up. Scientific regulations have also been made

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of untreated unruptured intracranial aneurysm (by CTA, MRA or DSA);
2. Patient with premorbid mRS of 3 or less;
3. Patient older than 14years;
4. Patient consenting to participate to the study;
5. Patients with a definite history of ischemic heart disease or ischemic stroke who accept antithrombotic or anticoagulant therapy for secondary pevention

Exclusion Criteria:

Subarachnoid hemorrhage with unknown causes;

- Page 4 of 4 [DRAFT] - 2. Patient with other cerebral arteriovenous malformations or cerebral arteriovenous fistulas; 3. Patient with malignant tumor; 4. Target aneurysm is fusiform, traumatic, mycotic, or dissecting related; 5. Inability to obtain informed consent; 6. Patients with a life expectancy less than 1 year; 7. Participating in the other clinical studies of intracranial aneurysm; 8. Refusal of follow-up

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients with unruptured intracranial aneurysms associated with ischemic heart disease or ischemic cerebrovascular disease,who accept antithrombotic or anticoagulant therapy
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Aneurysm rupture | Up to 4 years or time of aneurysm repair surgery
  Aneurysm rupture
Morphological changes of aneurysms | Up to 4 years or time of aneurysm repair surgery
  maximum diameter increase ≥ 1mm or appearance of a daughter sac

SECONDARY OUTCOMES:
Acute myocardial infarction | Up to 4 years]
  Acute myocardial infarction
New onset ischemic stroke | Up to 4 years]
  New onset ischemic stroke

CONTACTS AND LOCATIONS:
Overall Officials: Min He, M.D., Study Chair — West China Hospital

IPD SHARING:
Plan to Share IPD: No
share the original data 5 years after the study completion

REFERENCES:
- [Background] International Study of Unruptured Intracranial Aneurysms Investigators. Unruptured intracranial aneurysms--risk of rupture and risks of surgical intervention. N Engl J Med. 1998 Dec 10;339(24):1725-33. doi: 10.1056/NEJM199812103392401. PMID 9867550
- [Background] Wiebers DO, Whisnant JP, Huston J 3rd, Meissner I, Brown RD Jr, Piepgras DG, Forbes GS, Thielen K, Nichols D, O'Fallon WM, Peacock J, Jaeger L, Kassell NF, Kongable-Beckman GL, Torner JC; International Study of Unruptured Intracranial Aneurysms Investigators. Unruptured intracranial aneurysms: natural history, clinical outcome, and risks of surgical and endovascular treatment. Lancet. 2003 Jul 12;362(9378):103-10. doi: 10.1016/s0140-6736(03)13860-3. PMID 12867109
- [Background] UCAS Japan Investigators; Morita A, Kirino T, Hashi K, Aoki N, Fukuhara S, Hashimoto N, Nakayama T, Sakai M, Teramoto A, Tominari S, Yoshimoto T. The natural course of unruptured cerebral aneurysms in a Japanese cohort. N Engl J Med. 2012 Jun 28;366(26):2474-82. doi: 10.1056/NEJMoa1113260. PMID 22738097